CLINICAL TRIAL: NCT04837924
Title: The Effects of Fascia Iliaca Compartment Block on Hip Fracture Patients
Brief Title: Fascia Iliaca Compartment Block for Pain Management in Hip Fracture Patients
Acronym: BLOCKPAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital Sveti Duh (Other)
Responsible Party: Principal Investigator, Andela Simic, Principal Investigator, General Hospital Sveti Duh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0121812
Record Dates: First submitted 2021-03-24; First posted 2021-04-08 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Hip Fractures
Keywords: Hip Fractures; Pain Management
MeSH Terms: conditions — Hip Fractures; Agnosia | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: 80 participants, stratified randomization will be used, men/women, age 65-75 years/older then 75 years, The American Society of Anesthesiologists physical status classification, (ASA status) I-II/ ASA III and IV, and type of hip fracture intra/extracapsular
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be blinded by sham procedure (disinfection, sting with blunt needle, (without piercing the skin), in the groin area, same place where actual FICB is given and covered with same gauze/patch). It will not be revealed to care providers and outcome measurement associate in which group participant is. After the data collection statistical analyst will not know is A group experimental or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- B (FICB) (Experimental): Participants receiving fascia iliaca compartment block (FICB)
  Interventions: Procedure: fascia iliaca compartment block, (FICB) (levobupivacaine hydrochloride 0,25% 40 ml); Drug: paracetamol 1 gram IV; Drug: Rescue analgesic tramadol 100 mg IV if needed
- A (PLACEBO) (Sham Comparator): Participants receiving sham injection matching fascia iliaca compartment block (FICB)
  Interventions: Drug: paracetamol 1 gram IV; Drug: Rescue analgesic tramadol 100 mg IV if needed; Procedure: Sham injection

INTERVENTIONS:
Procedure: fascia iliaca compartment block, (FICB) (levobupivacaine hydrochloride 0,25% 40 ml) — Land mark technique will be used to perform FICB on the side of the hip fracture. The injection site is one centimetre caudal from the junction between medial 2/3 and lateral 1/3 in the imaginary line between anterior superior iliac spine and ipsilateral pubic tubercle. The goal is to administer local anesthetic in the fascia iliaca compartment.
  Arms: B (FICB)
Drug: paracetamol 1 gram IV — paracetamol 1 gram IV every six hours, 4 times in 24 hours
Drug: Rescue analgesic tramadol 100 mg IV if needed — Rescue analgesic, if needed, tramadol 100 mg in 100 ml saline (0,9% Sodium chloride) IV, up to 4 times in 24 hours
Procedure: Sham injection — Sting with blunt needle, (without piercing the skin), same site as fascia iliaca compartment block
  Arms: A (PLACEBO)

SUMMARY:
BLOCKPAIN is a randomized controlled study, 80 participants. The participants will be hip fracture patients in Emergency Medicine Department in Clinical Hospital "Sveti Duh", Zagreb, Croatia. Upon patient arrival inclusion and exclusion criteria will be established. After signing the informed consent form participant will be randomized in one of two study groups. One study group is fascia iliaca compartment block (FICB), the other is placebo. All participants will be given paracetamol 1 gram IV as standard care. If needed, rescue analgesic will be tramadol 100 mg in 100 ml saline IV. The time frame is 24 hours after the FICB or placebo procedure.

DETAILED DESCRIPTION:
Hip fractures in older patients are a major public health problem. For acute pain management, nonopioid analgesics are often not sufficient enough, and opioids have many adverse events. For this reasons fascia iliaca compartment block could be the treatment of choice. The objective of this study is to evaluate the efficacy of the fascia iliaca compartment block for pain management in the emergency department, especially the effect on stress response and the effect on the acute confusional state. The investigators intend to conduct a randomized clinical trial in hip fracture patients years 65 and older presenting in the emergency department. In addition to standard analgesia with parenteral paracetamol, the first group of patients will receive fascia iliaca compartment block and the second group placebo. The investigators will monitor the effect of treatment protocol on laboratory parameters of stress response copeptin and cortisol, frequency and severity of acute confusional state, pain intensity and the need for additional opioid analgesics. Data obtained from this research could significantly improve the standard and quality of analgesia in the older patients with hip fracture. Regional anesthesia can diminish or prevent the development of stress response and cognitive impairment and these are the factors that complicate recovery of this fragile group of patients.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture after minor trauma/simple falls, confirmed by imaging technique (X-ray or CT scan or MRI)
* signed informed consent form (after a verbal explanation and written information sheet)

Exclusion Criteria:

* pathological fracture
* head injury
* body mass bellow 50 kg
* cognitive impairment (Abbreviated Mental Test Score less then 6 points)
* oral anticoagulant drugs
* prior drug allergy (paracetamol, tramadol, local anesthetics)
* prior peripheral artery bypass surgery (on the same side as hip fracture)
* skin or soft tissue infection in the groin area (on the same side as hip fracture)
* simultaneously bilateral hip fracture
* opioid analgesics prior to hospital arrival

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Stress Response 1 | Change from baseline cortisol plasma level at 24 hours
  cortisol plasma level
Stress Response 2 | Change from baseline copeptin plasma level at 24 hours
  copeptin plasma level
Acute confusional state/Delirium | Change from baseline Abbreviated Mental Test Score at 24 hours
  Abbreviated Mental Test Score (AMTS) - 10 point scale, from 0 to 10, 10 is the best possible result, 2 and more point drop from baseline indicating delirium

SECONDARY OUTCOMES:
Pain Intensity | Immediately prior and 30, 120, 240 minutes and 24 hours
  Pain intensity at rest and pain intensity at movement, Numerical Rating Scale (NRS), from 0 to 10, 0 meaning "no pain" and 10 "the worst pain ever possible"

CONTACTS AND LOCATIONS:
Overall Officials: Anđela Simić, Principal Investigator — Clinical Hospital "Sveti Duh"
Locations (1):
- Clinical Hospital "Sveti Duh", Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared on demand, via Principal Investigator e-mail. There is a prior signed consent of all participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the study publication, unlimited
Access Criteria: The de-identified IPD will be available for research purposes by contacting the first author via e-mail.